CLINICAL TRIAL: NCT05263089
Title: Clinical Performance of Injectable Universal Flowable Composite Versus Conventional Resin Composite Restorations in Proximal Cavities of Posterior Teeth.
Brief Title: Clinical Performance of Injectable Universal Flowable Composite in Proximal Cavities of Posterior Teeth.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nanees Ayman Hassan Aly, Teaching Assistant, conservative Dentistry Department, Faculty of Dentistry, MSA university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Universal flowable composite
Record Dates: First submitted 2022-02-11; First posted 2022-03-02 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Proximal Cavities of Posterior Teeth
Keywords: Injectable universal flowable composite; Conventional resin composite; Randomized clinical trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Injectable Universal flowable resin composite
  Interventions: Other: PALFIQUE® Universal Flow; Tokuyama, Tokyo, Japan (super low flowability)
- Control (Active Comparator): Conventional resin composite
  Interventions: Other: ESTELITE® Alpha; Tokuyama, Tokyo, Japan

INTERVENTIONS:
Other: PALFIQUE® Universal Flow; Tokuyama, Tokyo, Japan (super low flowability) — Supplied in L-syringe with nozzle and dispensing Tips. "Super Low" has low flowability, non-slumping, non-running, and precision stacking properties. The layer dispensed will be 2 mm. in thickness and cured for 40 s.
  Other Names: Injectable Universal flowable resin composite
  Arms: Intervention
Other: ESTELITE® Alpha; Tokuyama, Tokyo, Japan — The composite was inserted using the incremental technique. Each increment of 2 mm was cured for 40 s.
  Other Names: Conventional resin composite
  Arms: Control

SUMMARY:
The aim of the study is to evaluate the clinical performance of injectable universal flowable composite vs conventional resin composite restorations in proximal cavities of posterior teeth. The null hypothesis is proposed that there will be no difference in the clinical performance of injectable universal flowable composite versus conventional resin composite restorations in proximal cavities of posterior teeth. The design for this randomized controlled clinical trial is a superiority framework with parallel groups with equal allocation ratios. The patients are randomly divided into two groups where one group will receive conventional resin composite and the other group will receive injectable universal flowable resin composite. The restorations will be evaluated for any fracture or loss of retention by using prob following Modified USPHS criteria at baseline, 3, 6, 12 month.

DETAILED DESCRIPTION:
The study will be conducted in the Conservative Dentistry Department, Faculty of Dentistry, Cairo University in conjunction with the Conservative Dentistry Department, Faculty of Dentistry, MSA University outpatient clinics. The predicted sample size was a total of 24. The sample size was increased by (20%) to account for possible dropouts during follow-up intervals to be total of (30) cases i.e. (15) for each group. Screening of patients that come to the Conservative Dentistry Department seeking dental care will continue until the target population is achieved. The patients will be subjected to examination and diagnosis. Once the patients that are potentially eligible for this study are identified, they will be contacted by the research operator who will explain the study and ascertain the patients' interest. If interested, more detailed evaluations and preparations, and schedule planning will be made. Then the patient will sign the informed consent to ensure the approval for all the prosecuted that will be done and his/her acceptance to participate in this trial. Randomization will be done using simple randomization by computerized sequence generation using www.random.org by generating numbers from 1:30 into two columns. Each participant will choose a random number from an opaque sealed envelope. When the participant chooses an envelope, it will be signed by the patient and the supervisor and the number on the envelope will be recorded in the patient chart to ensure that the patient is assigned to the randomized group. After anesthesia, prophylaxis was performed using a brush associated with pumice, mounted in a low-speed handpiece. The teeth will be cleaned from any plaque or debris. After shade selection, rubber dam isolation will be used to avoid any moisture contamination which might affect the clinical performance of the bond and restoration, and to provide favorable conditions for bond application, if any reason is found that contraindicate rubber dam usage the procedure will be done under the cotton roll and high suction insulation and the use of retraction cord if needed to avoid any moisture contamination. The class II preparations will be made with spherical diamond burs of appropriate size and removal of carious dentine will be performed with spherical carbide bur at low-speed hand-piece and hand instruments. The cavities were designed according to the principles of minimally invasive dentistry. The outline shape of the preparations will be limited to the removal of caries. No bevels were prepared. Minor finishing and polishing may be done to the teeth if needed to remove any sharp edges or friable/undermined enamel. PALFIQUE BOND (Palfique, Tokuyama, Japan) will be used with both types of resin composites to ensure standardization of the procedures. It is a one-component, one-coat application, self-etching, light-cured, dental adhesive system. By using the disposable applicator, the bond will be applied on the surface of the prepared cavity and then wait for 10 seconds or more. Then mild air is continuously applied to the surface for 5 seconds until the runny bond stays in the same position without any movement and light-cured for 10 seconds. Injectable Universal flowable resin composite (PALFIQUE® Universal Flow; Tokuyama, Tokyo, Japan) super-low flowability supplied in L-syringe with nozzle and dispensing Tips. "Super Low" has low flowability, non-slumping, non-running, and precision stacking properties. The layer dispensed will be 2 mm. in thickness and cured for 40 s. Conventional resin composite (ESTELITE® Alpha; Tokuyama, Tokyo, Japan). The composite was inserted using the incremental technique. Incremental filling techniques result in better light penetration and better polymerization of the composite resin, reduction of the cavity configuration factor, cuspal deflection, polymerization shrinkage stresses; and ensures that the resin adheres better to cavity walls. Each increment of 2 mm was cured for 40 s.

The restoration was performed for both groups using a pre-curved metallic sectional matrix, associated with a separating ring and a wooden wedge.

Following the removal of the matrix band, the proximal regions of the restorations were additionally polymerized buccally and lingually/palatally for 10 s.

Occlusal adjustments were made using articulating paper, and the quality of the interproximal contacts and cervical adaptation was checked by means of dental floss and interproximal radiographs. The restorations were finished with water-cooled fine and super-fine diamond burs. The polishing procedures of the occlusal surface were performed with abrasive rubber tips during the same appointment immediately after the restorative procedure for both groups. All participants will be instructed to follow oral hygiene measures to avoid plaque and bacterial accumulation which may negatively affect the clinical performance as fracture or loss of retention. The restoration will be evaluated for any fracture or loss of retention by using prob following Modified USPHS criteria.

ELIGIBILITY:
Participant Inclusion Criteria

* Adult patients aged 18-55 years.
* Patients with good oral hygiene (mild to moderate plaque accumulation).
* patients with asymptomatic compound proximal cavities in permanent posterior teeth.
* ICDAS (3 &4)

Teeth inclusion criteria

* Vital posterior teeth with compound proximal cavities.
* Teeth with no or minimum mobility
* No history of hypersensitivity in the teeth to be restored
* Free from signs and symptoms of pulpitis and pulpal necrosis.

Participant Exclusion criteria

* Patients who are unable to return for recall appointments.
* Patients with poor oral hygiene.
* Presence of abnormal oral, medical, or mental condition
* Patients with untreated extra occlusal stresses
* Patients with TMJ problems.

Teeth Exclusion criteria

* Root involvement.
* Periodontal disease that may affect the prognosis of the restoration or the tooth itself.
* Fractured or visibly cracked teeth.
* Presence of any developmental or formative defects.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-02 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Criteria of restoration evaluation indicating clinical performance. | 12 months
  The restoration will be evaluated for any fracture or loss of retention by using prob following Modified USPHS criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baroudi K, Rodrigues JC. Flowable Resin Composites: A Systematic Review and Clinical Considerations. J Clin Diagn Res. 2015 Jun;9(6):ZE18-24. doi: 10.7860/JCDR/2015/12294.6129. Epub 2015 Jun 1. PMID 26266238
- [Background] Bayraktar Y, Ercan E, Hamidi MM, Colak H. One-year clinical evaluation of different types of bulk-fill composites. J Investig Clin Dent. 2017 May;8(2). doi: 10.1111/jicd.12210. Epub 2016 Jan 22. PMID 26800647
- [Background] Ferracane JL, Lawson NC. Probing the hierarchy of evidence to identify the best strategy for placing class II dental composite restorations using current materials. J Esthet Restor Dent. 2021 Jan;33(1):39-50. doi: 10.1111/jerd.12686. Epub 2020 Nov 18. PMID 33206440
- [Background] Frascino S, Fagundes TC, Silva U, Rahal V, Barboza A, Santos PH, Briso A. Randomized Prospective Clinical Trial of Class II Restorations Using Low-shrinkage Flowable Resin Composite. Oper Dent. 2020 Jan/Feb;45(1):19-29. doi: 10.2341/18-230-C. Epub 2019 Apr 29. PMID 31034347
- [Background] Irmak O, Yaman BC, Orhan EO, Ozer F, Blatz MB. Effect of rubbing force magnitude on bond strength of universal adhesives applied in self-etch mode. Dent Mater J. 2018 Jan 30;37(1):139-145. doi: 10.4012/dmj.2017-018. Epub 2017 Oct 27. PMID 29081447
- [Background] Imai A, Takamizawa T, Sugimura R, Tsujimoto A, Ishii R, Kawazu M, Saito T, Miyazaki M. Interrelation among the handling, mechanical, and wear properties of the newly developed flowable resin composites. J Mech Behav Biomed Mater. 2019 Jan;89:72-80. doi: 10.1016/j.jmbbm.2018.09.019. Epub 2018 Sep 17. PMID 30265868
- [Background] Ikeda I, Otsuki M, Sadr A, Nomura T, Kishikawa R, Tagami J. Effect of filler content of flowable composites on resin-cavity interface. Dent Mater J. 2009 Nov;28(6):679-85. doi: 10.4012/dmj.28.679. PMID 20019418
- [Background] Jang JH, Park SH, Hwang IN. Polymerization shrinkage and depth of cure of bulk-fill resin composites and highly filled flowable resin. Oper Dent. 2015 Mar-Apr;40(2):172-80. doi: 10.2341/13-307-L. Epub 2014 Aug 19. PMID 25136904
- [Background] Kramer N, Reinelt C, Frankenberger R. Ten-year Clinical Performance of Posterior Resin Composite Restorations. J Adhes Dent. 2015 Aug;17(5):433-41. doi: 10.3290/j.jad.a35010. PMID 26525008
- [Background] Kitasako Y, Sadr A, Burrow MF, Tagami J. Thirty-six month clinical evaluation of a highly filled flowable composite for direct posterior restorations. Aust Dent J. 2016 Sep;61(3):366-73. doi: 10.1111/adj.12387. PMID 26573239
- [Background] Lai G, Zhao L, Wang J, Kunzelmann KH. Surface properties and color stability of dental flowable composites influenced by simulated toothbrushing. Dent Mater J. 2018 Sep 30;37(5):717-724. doi: 10.4012/dmj.2017-233. Epub 2018 Jul 12. PMID 29998939
- [Background] Loguercio AD, Luque-Martinez I, Lisboa AH, Higashi C, Queiroz VA, Rego RO, Reis A. Influence of Isolation Method of the Operative Field on Gingival Damage, Patients' Preference, and Restoration Retention in Noncarious Cervical Lesions. Oper Dent. 2015 Nov-Dec;40(6):581-93. doi: 10.2341/14-089-C. Epub 2015 Jul 9. PMID 26158415
- [Background] Stape THS, Wik P, Mutluay MM, Al-Ani AAS, Tezvergil-Mutluay A. Selective dentin etching: A potential method to improve bonding effectiveness of universal adhesives. J Mech Behav Biomed Mater. 2018 Oct;86:14-22. doi: 10.1016/j.jmbbm.2018.06.015. Epub 2018 Jun 8. PMID 29913306
- [Background] Shaalan OO, Abou-Auf E, El Zoghby AF. Clinical evaluation of flowable resin composite versus conventional resin composite in carious and noncarious lesions: Systematic review and meta-analysis. J Conserv Dent. 2017 Nov-Dec;20(6):380-385. doi: 10.4103/JCD.JCD_226_17. PMID 29430087
- [Background] Stefanski S, van Dijken JW. Clinical performance of a nanofilled resin composite with and without an intermediary layer of flowable composite: a 2-year evaluation. Clin Oral Investig. 2012 Feb;16(1):147-53. doi: 10.1007/s00784-010-0485-8. Epub 2010 Nov 23. PMID 21104100
- [Background] Sumino N, Tsubota K, Takamizawa T, Shiratsuchi K, Miyazaki M, Latta MA. Comparison of the wear and flexural characteristics of flowable resin composites for posterior lesions. Acta Odontol Scand. 2013 May-Jul;71(3-4):820-7. doi: 10.3109/00016357.2012.734405. PMID 23638859
- [Background] Rocha Gomes Torres C, Rego HM, Perote LC, Santos LF, Kamozaki MB, Gutierrez NC, Di Nicolo R, Borges AB. A split-mouth randomized clinical trial of conventional and heavy flowable composites in class II restorations. J Dent. 2014 Jul;42(7):793-9. doi: 10.1016/j.jdent.2014.04.009. Epub 2014 Apr 25. PMID 24769385
- [Background] van Dijken JW, Pallesen U. A six-year prospective randomized study of a nano-hybrid and a conventional hybrid resin composite in Class II restorations. Dent Mater. 2013 Feb;29(2):191-8. doi: 10.1016/j.dental.2012.08.013. Epub 2012 Oct 9. PMID 23063254
- [Background] Veloso SRM, Lemos CAA, de Moraes SLD, do Egito Vasconcelos BC, Pellizzer EP, de Melo Monteiro GQ. Clinical performance of bulk-fill and conventional resin composite restorations in posterior teeth: a systematic review and meta-analysis. Clin Oral Investig. 2019 Jan;23(1):221-233. doi: 10.1007/s00784-018-2429-7. Epub 2018 Mar 28. PMID 29594349
- [Background] Wang Y, Li C, Yuan H, Wong MC, Zou J, Shi Z, Zhou X. Rubber dam isolation for restorative treatment in dental patients. Cochrane Database Syst Rev. 2016 Sep 20;9(9):CD009858. doi: 10.1002/14651858.CD009858.pub2. PMID 27648846
- [Background] Yazici AR, Kutuk ZB, Ergin E, Karahan S, Antonson SA. Six-year clinical evaluation of bulk-fill and nanofill resin composite restorations. Clin Oral Investig. 2022 Jan;26(1):417-426. doi: 10.1007/s00784-021-04015-2. Epub 2021 Jun 10. PMID 34110494